CLINICAL TRIAL: NCT06640530
Title: A Double-Blind, Randomized Clinical Study of the Efficacy and Safety of BCD-263 and Opdivo® as Monotherapy in Subjects With Advanced Melanoma of the Skin
Brief Title: Clinical Study of the Efficacy and Safety of BCD-263 and Opdivo® as Monotherapy in Subjects With Advanced Melanoma of the Skin
Acronym: UNIVERSE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-263-2
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma; Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCD-263 (Experimental): BCD-263 will be administered during main period and open-label period
  Interventions: Drug: BCD-263
- Opdivo (Active Comparator): Opdivo will be administered during main period
  Interventions: Drug: Opdivo

INTERVENTIONS:
Drug: BCD-263 — BCD-263 at a dose 480 mg administered intravenously every 4 weeks up to 6 cycles
  Other Names: Nivolumab
  Arms: BCD-263
Drug: Opdivo — Opdivo at a dose 480 mg administered intravenously every 4 weeks up to 6 cycles
  Other Names: Nivolumab
  Arms: Opdivo

SUMMARY:
The aim of the study BCD-263-2/UNIVERSE is to demonstrate comparable efficacy and similar safety and immunogenicity profile of BCD-263 and Opdivo after repeated intravenous doses in subjects with advanced unresectable or metastatic melanoma of the skin.

DETAILED DESCRIPTION:
Following screening, subjects will be randomized to receive either BCD-263 or Opdivo in a 1:1 ratio and enter the main study period.

During the main study period, subjects will receive therapy with BCD-263 or Opdivo, which will be administered intravenously until disease progression or signs of unacceptable toxicity develop (whichever occurs earlier).

At Week 25, after completion of all scheduled procedures subjects in both groups will continue to receive open-label BCD-263 for up to a total of 2 years of therapy, or disease progression, or signs of unacceptable toxicity (whichever occurs first).

Following discontinuation of the study therapy, the subjects will enter a follow-up period, during which data on overall survival will be collected through telephone contacts.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and the subject's ability to comply with the protocol requirements.
2. Age ≥18 years at the time of signing the informed consent form.
3. Histologically confirmed melanoma with the following prognostic characteristics:

   * LDH <ULN of local laboratory (enrollment of subjects with LDH <2 x ULN of local laboratory is allowed until the number of subjects with LDH >ULN is 30% of the total population of randomized subjects. The Sponsor will inform when enrollment of subjects is limited by LDH level <ULN of the local laboratory).
   * Absence, according to the Investigator, of clinically significant symptoms associated with the tumor.
   * Absence, according to the Investigator, of rapidly progressing metastatic melanoma.
4. Newly diagnosed advanced unresectable (stage III) or metastatic disease (stage IV), or progressive disease during / relapsing after radical treatment.
5. Presence of a tumor sample (archived or new biopsy) that is suitable for evaluation for PD L1 expression in the Investigator's opinion.
6. At least one measurable lesion as per RECIST 1.1 based on independent central review.
7. ECOG score 0-1.
8. Laboratory test results consistent with adequate functioning of systems and organs.

Exclusion Criteria:

1. Indications for radical treatment (surgery, radiation therapy).
2. Uveal or mucosal melanoma.
3. Previous systemic anticancer therapy for advanced unresectable or metastatic skin melanoma.
4. Active CNS metastases and/or carcinomatous meningitis.
5. Previous invasive cancer, excluding diseases treated with potentially radical therapy with no evidence of recurrence for 2 years from the start of this therapy (subjects with radically resected basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ of the uterus and other carcinomas in situ may be included).
6. Subjects with severe concomitant disorders, life-threatening acute complications of the primary disease (including massive pleural, pericardial, or peritoneal effusions requiring intervention, pulmonary lymphangitis, bleeding or organ perforation) at the time of signing the informed consent and during the screening period.
7. Concomitant diseases and/or conditions that significantly increase the risk of adverse events (AEs) during the study.
8. Active, known or suspected autoimmune disorders (subjects with type 1 diabetes mellitus or hypothyroidism requiring only hormone-replacement therapy and those with skin disorders [vitiligo, alopecia, or psoriasis] not requiring systemic therapy are eligible to participate).
9. The need for systemic corticosteroids (at doses equivalent to >10 mg/day prednisolone) or any other immunosuppressive drugs within 14 days prior to randomization. The use of inhaled and topical corticosteroids is allowed.
10. History of (non-infectious) pneumonitis requiring corticosteroid therapy or pneumonitis at the time of screening.
11. Any anticancer therapy or major surgery within 28 days prior to randomization, or the subject's AE (other than alopecia) caused by anticancer therapy has not yet recovered to CTCAE grade 1 or has not completely resolved.
12. Concomitant use of drugs or medical devices studied in other clinical studies or their use within 28 days prior to randomization.
13. Infections requiring therapy or systemic antibiotics within 14 days prior to randomization.
14. Administration of a live and/or attenuated vaccine within 28 days prior to randomization.
15. Positive HIV-1 or HIV-2 test.
16. HBV/HCV infections (subjects with a negative PCR result for hepatitis C virus RNA, without significant abnormalities in blood chemistry tests, examined by an infectious disease specialist and not requiring specific antiviral treatment at the time of screening, may be included in the study. Subjects with a positive HbsAg test result cannot be included in the study).
17. Impossibility to administer intravenous contrast agents (including due to hypersensitivity to contrast media).
18. Hypersensitivity or allergy to any of the nivolumab product components. Hypersensitivity or allergy to medicinal products obtained based on Chinese hamster ovary cells, or history of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or hybrid proteins.
19. Pregnancy or breastfeeding, as well as intention to become pregnant or father a child during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) according to RECIST 1.1 | Week 25
  To compare the overall response rates (ORRs) after administration of BCD-263 and Opdivo in subjects with advanced unresectable or metastatic skin melanoma

SECONDARY OUTCOMES:
Time to response | Week 25
  To compare time to response according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Duration of response | week 25
  To compare duration of response according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
DCR | week 25
  To compare disease control rate according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
PFS | week 25
  To compare progression-free survival according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Overall survival | week 25
  To compare overall survival according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Safety assessment | Through week 105
  The subjects will undergo the vital sign assessment, physical and instrumental examination, sampling for complete blood count, blood chemistry, thyroid hormone tests, and urinalysis, as well as assessment of the presence and characteristics of adverse events to assess the safety of the investigational product
Immunogenicity assessment | Through week 105
  Proportion of subjects with binding and/or neutralizing antibodies to nivolumab

OTHER OUTCOMES:
AUC(0-∞) (optional) | week 25
  To compare area under the drug concentration-time curve in the time interval from 0 to ∞ after intravenous administration of BCD-263 and Opdivo
AUC(0-672) of nivolumab (optional) | week 25
  To compare area under the drug concentration-time curve in the time interval from 0 to 672 hours after intravenous administration of BCD-263 and Opdivo
Cmax (optional) | week 25
  To compare the maximum concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
Tmax (optional) | week 25
  To compare time to the maximum concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
T½ (optional) | week 25
  To compare half-life period of nivolumab after intravenous administration of BCD-263 and Opdivo
Kel (optional) | week 25
  To compare elimination rate constant of nivolumab after intravenous administration of BCD-263 and Opdivo
Vd (optional) | week 25
  To compare steady-state volume of distribution of nivolumab after intravenous administration of BCD-263 and Opdivo
Cl (optional) | week 25
  To compare total clearance of nivolumab after intravenous administration of BCD-263 and Opdivo
Ceoi (optional) | week 25
  To compare plasma concentration at the and of infusion of nivolumab after intravenous administration of BCD-263 and Opdivo
Cmin (optional) | week 25
  To compare minimal concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
Cmax, ss (optional) | week 25
  To compare steady-state maximum concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
Ctrough, ss (optional) | week 25
  To compare steady-state trough concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
Ctrough (optional) | week 25
  To compare trough concentration of nivolumab after intravenous administration of BCD-263 and Opdivo

CONTACTS AND LOCATIONS:
Locations (44):
- Belarus (4):
  - Healthcare Institution "Brest Regional Oncological Dispensary", Brest
  - Health Institution "Gomel Regional Clinical Oncology Center", Homyel
  - Healthcare Institution "Minsk City Clinical Cancer Center", Minsk
  - State Institution "Republic Scientific and Practical Centre for Oncology and Medical Radiology Named after N.N.Aleksandrov", Minsk
- Pakistan (2):
  - Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad
  - Rehman Medical Institute, Peshawar
- Russia (38):
  - Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine, Chelyabinsk, Chelyabinsk Oblast
  - Clinical Oncologic Dispensary No. 1, Krasnodar, Krasnodar Kari
  - Krasnoyarsk Regional Clinical Oncological Dispensary named after A.I. Kryzhanovsky, Krasnoyarsk, Krasnoyarsk Krai
  - JSC "Modern Medical Technologies", Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg, Sankt-Peterburg
  - State Budgetary Institution of Healthcare of the Arkhangelsk Region "Severodvinsk City Hospital №2 of Emergency", Arkhangelsk
  - Regional State Budgetary Healthcare Institution "Altai Regional Oncological Dispensary", Barnaul
  - Ivanovo Regional Oncology Center, Ivanovo
  - State Health Care Institution "Republican Clinical Cancer Center," the Ministry of Health of the Udmurt Republic, Izhevsk
  - State Budgetary Health Institution "Regional Clinical Hospital of Kaliningrad Region", Kaliningrad
  - State Budgetary Healthcare Institution of Kaluga Region "Kaluga Region Clinical Oncological Dispensary", Kaluga
  - State Autonomous Health Institution "Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor M.Z. Sigal", Kazan'
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - JSC "Medsi Group", Moscow
  - Moscow City Oncology Hospital No. 62, Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Oncology Hospital No. 1 of the Department of Health of the City of Moscow", Moscow
  - State Budgetary Healthcare Institution "Moscow Clinical Scientific Center funded by Moscow Health Department" (SBHI MCSC MHD), Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "Moscow Multidisciplinary Clinical Center "Kommunarka" of the Department of Health of the City of Moscow", Moscow
  - Nizhny Novgorod Region State Budgetary Healthcare Institution "Nizhny Novgorod Regional Clinical Oncological Dispensary", Nizhny Novgorod
  - State Budgetary Healthcare Institution "Novosibirsk Regional Clinical Oncology Center" of the Novosibirsk Region, Novosibirsk
  - State budget healthcare institution Omsk region "Clinical Oncology Dispensary", Omsk
  - Perm Region Oncology Dispensary, Perm
  - State Budgetary Healthcare Institution of Perm Krai "Order of Honour" Perm Regional Clinical Hospital ", Perm
  - Federal Government Budgetary Institution "National Institute of Cancer Research" of Ministry of Health of Russian Federation, Rostov-on-Don
  - Private healthcare institution "Clinical hospital "RZD-Medicine" of the city of Saint Petersburg", Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov Research Institute of Oncology" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - JSC "North-West Centre of Evidence-Based Mediccine", Saint Petersburg
  - Limited Liability Company "Oncological Research Center", Saint Petersburg
  - Private Medical Institution Evromedservis, Saint Petersburg
  - State-financed Health Institution "Samara Region Clinical Oncology Dispensary", Samara
  - Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva ", Saransk
  - Provincial health official body "Smolensk Regional Clinical Oncological Dispensary", Smolensk
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University" of the Ministry of Health of the Russian Federation, Tomsk
  - Federal State Budgetary Institution of Health "Tver Regional Clinical Oncological Dispensary" of the Tver Region, Tver'
  - State Autonomus Institution of Health "Mulitiprofile Clinical Medical Centre "Medical City"", Tyumen
  - Republican Clinical Oncology Dispensary of Ministry of Health republic Bashkortostan, Ufa
  - State Health Care Institution "Volgograd Regional Clinical Oncology Dispensary № 1", Volgograd
  - Sverdlovsk Regional Oncology Center, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No